CLINICAL TRIAL: NCT06808399
Title: Lower Limb Functional Asymmetry in Healthy Novice, Moderately and Highly-trained Distance Runners Versus Non-athletes
Brief Title: The Magnitude of Inter-limb Asymmetry and Its Assocation with Inter-limb Asymmetry in Distance Runners and Non-runners
Acronym: ASYMRUN
Status: Recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Joachim D'Hondt, PhD Researcher, Vrije Universiteit Brussel
Other Study IDs: 22381Asymrun
Record Dates: First submitted 2022-11-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Highly-trained distance runners: This study is an observational study and not an interventional study.
- Novice distance runners: This study is an observational study and not an interventional study.
- Non-Athletes: This study is an observational study and not an interventional study.
- Moderately trained distance runners: This study is an observational study and not an interventional stud

SUMMARY:
Distance running is one of the most popular and most accessible ways to engage in physical activity. Although distance running offers numerous health-related benefits and protects against noncommunicable diseases (e.g., type 2 diabetic, obesity, hypertension), research has indicated a high prevalence of running-related injuries with a more pronounced incidence among novice runners (i.e., 17.8 injuries per 1000h) compared to their highly trained peers (i.e., 7.2 injuries per 1000h).

Interlimb asymmetry has previously been related to higher injury risk as well as to impaired sports performances. Nevertheless, to date, research on the degree and evolution of functional asymmetry (e.g., unequal strength between limbs) in distance runners is scarce and the role of functional asymmetries in running performance and running-related injuries remains unclear. Moreover, and despite the great number of unilateral tests available in the literature, there currently exists no reliable and run-specific field-based test battery to examine the degree of lower limb asymmetry in distance runners. Therefore, this study aims to assess the test-retest, intra- and inter-rater reliability of a newly created running-specific field-based test battery to assess the presence and degree of functional lower limb asymmetry among novice, moderatly and highly trained distance runners as well as a control group of non-athletes. The second objective is to assess the association between inter-limb asymmetry and running performance.

ELIGIBILITY:
Inclusion Criteria:

* • Being aged between 20 and 50 years at Tfamiliarization

  * Being free from any medical attention injury (i.e., injury that results in a participant receiving medical attention) for at least 6 months upon Tfamiliarization
  * Speaking Dutch, French or English
* Highly trained distance runners:

  * Running at least 150km per month for at least 3 months

Moderately-trained runners:

* Running between 40 - 150 km per month for at least 6 months

  - Novice distance runners:
* Running not more than 10km per week for the past 12 months

  - Control group of non-athletes
* Performing <75min of systematic moderate to vigorous-intensity physical activity per week and having no experience in systematic (un)structured running activities for the past 5 years

Exclusion Criteria:

* • Being younger than 20 years or older than 50 years at Tfamiliarization

  * Any known relevant medical history or current condition (e.g., neurological diseases, inner ear diseases) that could affect the performance of the functional tests (e.g., balance in repeated hop tests)
  * Participants that have undergone a surgery at lower limb level during the past 6 months
  * Medication or drug use (e.g., blood pressure medicines)that could affect the performance of the functional tests (e.g., balance in repeated hop tests)
  * Participants performing more than two hours per week of unilateral sports (e.g., tennis or soccer)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy population (see eligibility criteria)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Lean mass | Baseline
  Measured using dual-energy X-ray absorptiometry.
Fat mass | Baseline
  Measured using dual-energy X-ray absorptiometry.
Bone mineral density | Baseline
  Measured using dual-energy X-ray absorptiometry.
Phase angle | Baseline
  Measured using bioelectrical impedance analysis.
Lean mass | Baseline
  Measured using bioelectrical impedance analysis.
Fat mass | Baseline
  Measured using bioelectrical impedance analysis.
Total segmental water | Baseline
  Measured using bioelectrical impedance analysis.
Extracellular water | Baseline
  Measured using bioelectrical impedance analysis.
5 repeated vertical hop test. | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using an Optojump device
5 repeated horizontal hop test | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using an Optojump device
ankle dorsiflexion range of motion | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  The maximal dorsiflexion range of motion (cm from a wall) will be measured with tape measure.
Side bridge endurance test | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  The side bridge endurance test will be carried out in which, the participants will lie on one side of the body fully extended (i.e., hip and torso at 0°) in a plank position with the feet elevated on a 15-cm step and with the superior feet placed in front. The participants will be instructed to lift the hips until the body is in straight position with the arms folded across the chest. The time until a drop (lasting more than 3s) of the hips from the optimal position will manually be recorded. To control for a full range of motion upon the execution of this muscle capacity tests, a reference dowel will be used to indiciate the desired range of motion.
Hip adduction strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured with a handheld dynamometer.
Hip abduction strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using a hand-held dynamometer.
Knee extension strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using a hand-held dynamometer.
Knee flexion strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using a hand-held dynamometer.
Ankle dorsiflexion strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using a hand-held dynamometer.
Ankle plantar flexion strength | 3 test occasions: baseline, 2 weeks after baseline and 4 weeks after baseline.
  Measured using a hand-held dynamometer.
Cooper test | This test will be carried out on the second test occasion (two weeks after baseline).
  Maximal distance covered in 12 minutes.
Training volume | Baseline
  Surveyed with an online questionnaire and quantified in hours/week (per sport performed).
Contact time while running | This test will be carried out on the third test occasion (four weeks after baseline).
  Measures with an Optojump device
Flight time while running | This test will be carried out on the third test occasion (four weeks after baseline).
  Measured using an Optojump device.
Stride length | This test will be carried out on the third test occasion (four weeks after baseline).
  Measured using an Optojump device.

SECONDARY OUTCOMES:
Weight | Baseline
Height | Baseline
Leg length | Baseline
  Measured using dual-energy X-ray absorptiometry and a tape measure.
Bone mineral content | Baseline
  Measured busing dual-energy X-ray absorptiometry.

CONTACTS AND LOCATIONS:
Locations (1):
- MOVE Research group, Ixelles-Elsene, Brussels Capital, Belgium